CLINICAL TRIAL: NCT02527200
Title: Effect of Liraglutide for Weight Management in Paediatric Subjects With Prader-Willi Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-4179; 2014-004415-37 (EudraCT Number); U1111-1162-7884 (Other: WHO); NL54145.078.15 (Other: CCMO)
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Injected s.c./ subcutaneously (under the skin) This trial consists of a part A and a part B. Part A of the trial is conducted in obese adolescents with PWS. Part B of the trial is conducted in obese children with PWS. Entry into part A and part B of the trial will be sequential.
  Arms: Liraglutide
Drug: placebo — Injected s.c./ subcutaneously (under the skin) This trial consists of a part A and a part B. Part A of the trial is conducted in obese adolescents with PWS. Part B of the trial is conducted in obese children with PWS. Entry into part A and part B of the trial will be sequential.
  Arms: Placebo

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate the effect of liraglutide for weight management in paediatric subjects with Prader-Willi Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Confirmed diagnosis of PWS (Prader-Willi Syndrome) (by genetic testing)
* Male or female, age at the time of signing informed consent: - Part A: above or equal to 12 years and less than 18 years
* Tanner stage 2-5 pubertal development for part A, and Tanner stage 1 for part B
* BMI (body mass index) corresponding to equal or above 30 kg/m^2 for adults by international cut-off points1 and equal or above the 95th percentile for age and sex (for diagnosis of obesity)
* Stable body weight during the previous 90 days before screening ( below 10 kg self-reported weight change)
* Testing has been performed to evaluate for adrenal insufficiency and documented in medical record

Exclusion Criteria:

* Type 1 diabetes mellitus (T1DM)
* Type 2 diabetes mellitus (T2DM)
* Calcitonin equal or above 50 ng/L
* No change in treatment plan with growth hormone (GH) from randomisation to the end of the open-label period patients on growth hormone to stay on, patients off GH to stay off during this period. Adjustments in doses of growth hormone will be permitted)
* Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN2) or Medullary Thyroids Carcinoma (MTC)
* History of pancreatitis (acute or chronic)
* Treatment with any medication prescribed for weight loss within 90 days before screening (e.g. orlistat, zonisamide, topiramate/phentermine, lorcaserin, phentermine, bupropion/naltrexone,liraglutide, metformin)
* Untreated adrenal insufficiency
* Suggestive history of, or significant risk of gastroparesis (e.g. marked abdominal bloating post meal, history of vomiting, severe constipation), as judged by the Investigator

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (5):
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, Columbus, Ohio
- Australia (2):
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, Parkville, Victoria
- Canada (2):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Montreal, Quebec
- France (12):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Bordeaux
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Haguenau
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Marseille Cédex 05
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Nice
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Rouen
  - Novo Nordisk Investigational Site, Toulouse
- Italy (3):
  - Novo Nordisk Investigational Site, Fiumicino
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Padua
- Novo Nordisk Investigational Site, Rotterdam, Netherlands
- Novo Nordisk Investigational Site, Grafton, New Zealand
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Samsun
  - Novo Nordisk Investigational Site, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
According to Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Diene G, Angulo M, Hale PM, Jepsen CH, Hofman PL, Hokken-Koelega A, Ramesh C, Turan S, Tauber M. Liraglutide for Weight Management in Children and Adolescents With Prader-Willi Syndrome and Obesity. J Clin Endocrinol Metab. 2022 Dec 17;108(1):4-12. doi: 10.1210/clinem/dgac549. PMID 36181471
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 20 sites in 8 countries as follows: Australia (2), Canada (1), France (7), Italy (2), Netherlands (1), New Zealand (1), Turkey (3), and the United States (3).
Pre-assignment Details: Trial has part A & B, participants entered sequentially into part A & B, and were randomised 2:1 (liraglutide/placebo). Part A conducted in adolescents (≥12-<18 years [yrs], Tanner stage 2-5) with Prader-Willi Syndrome (PWS) and obesity; Part B in children (≥6-˂12 yrs, Tanner stage below 2 with PWS and obesity. On part A 16-week double-blind period completion, data monitoring committee reviewed PK data to un-blind part A safety data then recommended randomisation (liraglutide/placebo) in part B.
Groups:
- Part A: Liraglutide: Participants received once daily subcutaneous injection of liraglutide for 52 weeks. Dosing was initiated with liraglutide 0.6 mg daily for one week and increased in weekly dosage steps of 0.6 mg until a maximum tolerated dose (MTD) (as judged by the Investigator) or a dose of 3.0 mg liraglutide was reached, i.e., 0.6 mg (week 1), 1.2 mg (week 2), 1.8 mg (week 3), 2.4 mg (week 4) and 3.0 mg (week 5 to week 52).
- Part A: Placebo; Part B: Placebo: Participants received once daily subcutaneous injection of placebo matched to liraglutide for 16 weeks.
- Part B: Liraglutide: Participants received once daily subcutaneous injection of liraglutide for 52 weeks. For children with body weight ≥ 45 kg; dosing was initiated with liraglutide 0.6 mg daily for one week and increased in weekly dosage steps of 0.6 mg until a MTD (as judged by the Investigator) or a dose of 3.0 mg liraglutide was reached, i.e., 0.6 mg (week 1), 1.2 mg (week 2), 1.8 mg (week 3), 2.4 mg (week 4) and 3.0 mg (week 5 to week 52). For children with body weight <45 kg: dosing was initiated with liraglutide 0.3 mg daily for one week and increased to 0.6 mg after the first week. Thereafter, the dose was increased in weekly steps of 0.6 mg until an MTD (as judged by the Investigator) or a dose of 2.4 mg liraglutide was reached. i.e., 0.3 mg (week 1), 0.6 mg (week 2), 1.2 mg (week 3), 1.8 mg (week 4), 2.4 mg (week 5 to week 52).
Period: Overall Study
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo
Started | 20 | 12 | 17 | 7
Safety Analysis Set (SAS) | 20 | 12 | 17 | 7
Full Analysis Set (FAS) | 19 | 12 | 17 | 7
Completed | 17 | 9 | 15 | 7
Not Completed | 3 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 0
Not completed — Unclassified | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) which included all randomised participants who received at least one dose of trial product and had any post-randomisation data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Total
Number analyzed (Participants) | 19 | 12 | 17 | 7 | 55
Age, Customized [Count of Participants; unit: Participants]
  6 - <12 years | 0 | 0 | 17 | 7 | 24
  12 - <18 years | 19 | 12 | 0 | 0 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 11 | 2 | 28
  Male | 9 | 7 | 6 | 5 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 1 | 5
  Not Hispanic or Latino | 18 | 12 | 11 | 6 | 47
  Unknown or Not Reported | 0 | 0 | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 0 | 1 | 0 | 3
  White | 11 | 6 | 10 | 7 | 34
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 5 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index (BMI) Standard Deviation Score (SDS) From Baseline to 16 Weeks
Description: Change in BMI SDS from baseline to week 16 is presented. BMI SDS also called Z-scores, was calculated using the following formula: Z=[(y / M)^L - 1] / S*L; where L, M and S are median (M), Box-cox power (L) and variation coefficient (S) of children/adolescents', y= individual BMI. BMI provided for each sex and age. For each participant, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. Possible values range from -3 to +3, a negative score being beneficial.
Time Frame: Week 0, Week 16
Population: Full analysis set (FAS) which included all randomised participants who received at least one dose of trial product and had any post-randomisation data. Overall Number of Participants Analyzed" = number of participants who contributed to the analysis. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Mean (Standard Deviation); unit: SDS score
Groups:
- Part A+B: Liraglutide: Participants received once daily subcutaneous (under the skin) injection of liraglutide for 52 weeks (open label for 16 weeks and double-blinded for 36 weeks ) in a dose escalating manner. For both part A and part B (for children with body weight ≥ 45 kilograms (kg)): dosing was initiated with liraglutide 0.6 milligrams (mg) daily for one week and increased in weekly dosage steps of 0.6 mg until a maximum tolerated dose (MTD) (as judged by the Investigator) or a dose of 3.0 mg liraglutide was reached, i.e., 0.6 mg (week 1), 1.2 mg (week 2), 1.8 mg (week 3), 2.4 mg (week 4) and 3.0 mg (week 5 to week 52). For Part B children with body weight < 45 kg: dosing was initiated with liraglutide 0.3 mg daily for one week and increased to 0.6 mg after the first week. Thereafter, the dose was increased in weekly steps of 0.6 mg until an MTD (as judged by the Investigator) or a dose of 2.4 mg liraglutide was reached. i.e., 0.3 mg (week 1), 0.6 mg (week 2), 1.2 mg (week 3), 1.8 mg (week 4), 2.4 mg (week 5 to week 52).
- Part A+B: Placebo: Participants received once daily subcutaneous injection of placebo matched to liraglutide for 16 weeks (open label).
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 16 | 7 | 34 | 19
SDS score | -0.18 (0.21) | -0.18 (0.23) | -0.50 (0.65) | -0.48 (0.39) | -0.33 (0.49) | -0.29 (0.32)

2. Primary Outcome: Change in Body Mass Index (BMI) Standard Deviation Score (SDS) From Baseline to 52 Weeks
Description: Change in BMI SDS from baseline to week 52 is presented. BMI SDS also called Z-scores, was calculated using the following formula: Z=[(y / M)^L - 1] / S*L; where L, M and S are median (M), Box-cox power (L) and variation coefficient (S) of children/adolescents', y= individual BMI. BMI provided for each sex and age. For each participant, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. Possible values range from -3 to +3, a negative score being beneficial.
Time Frame: Week 0, Week 52
Population: FAS which included all randomised participants who received at least one dose of trial product and had any post-randomisation data. Overall Number of Participants Analyzed = number of participants who contributed to the analysis. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 14 | 7 | 31 | 18
SDS score | -0.27 (0.37) | -0.13 (0.25) | -0.79 (1.21) | -0.71 (0.68) | -0.50 (0.88) | -0.36 (0.53)

3. Secondary Outcome: Percentage of Participants Achieving ≥ 5% Reduction in Baseline BMI at Week 16
Description: Percentage of participants achieving more than or equal to (≥) 5% reduction in their baseline (week 0) BMI at week 16 is presented. In below table, 'Yes' infers percentage of participants who achieved ≥ 5% reduction in their baseline (week 0) BMI at week 16 and 'No' infers percentage of participants who did not achieve ≥ 5% reduction in their baseline (week 0) BMI at week 16.
Time Frame: At week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 16 | 7 | 34 | 19
Percentage of participants
  Yes | 27.8 | 8.3 | 37.5 | 57.1 | 32.4 | 26.3
  No | 72.2 | 91.7 | 62.5 | 42.9 | 67.6 | 73.7

4. Secondary Outcome: Percentage of Participants Achieving ≥ 5% Reduction in Baseline BMI at Week 52
Description: Percentage of participants achieving more than or equal to (≥) 5% reduction in their baseline (week 0) BMI at week 52 is presented. In below table, 'Yes' infers percentage of participants who achieved ≥ 5% reduction in their baseline (week 0) BMI at week 52 and 'No' infers percentage of participants who did not achieve ≥ 5% reduction in their baseline (week 0) BMI at week 52.
Time Frame: At week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 14 | 7 | 31 | 18
Percentage of participants
  Yes | 29.4 | 18.2 | 35.7 | 42.9 | 32.3 | 27.8
  No | 70.6 | 81.8 | 64.3 | 57.1 | 67.7 | 72.2

5. Secondary Outcome: Percentage of Participants Achieving ≥ 10% Reduction in Baseline BMI at Week 16
Description: Percentage of participants achieving more than or equal to (≥) 10% reduction in their baseline (week 0) BMI at week 16 is presented. In below table, 'Yes' infers percentage of participants who achieved ≥ 10% reduction in their baseline (week 0) BMI at week 16 and 'No' infers percentage of participants who did not achieve ≥ 10% reduction in their baseline (week 0) BMI at week 16.
Time Frame: At week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 16 | 7 | 34 | 19
Percentage of participants
  Yes | 0 | 0 | 6.3 | 14.3 | 2.9 | 5.3
  No | 100 | 100 | 93.8 | 85.7 | 97.1 | 94.7

6. Secondary Outcome: Percentage of Participants Achieving ≥ 10% Reduction in Baseline BMI at Week 52
Description: Percentage of participants achieving more than or equal to (≥) 10% reduction in their baseline (week 0) BMI at week 52 is presented. In below table, 'Yes' infers percentage of participants who achieved ≥ 10% reduction in their baseline (week 0) BMI at week 52 and 'No' infers percentage of participants who did not achieve ≥ 10% reduction in their baseline (week 0) BMI at week 52.
Time Frame: At week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 14 | 7 | 31 | 18
Percentage of participants
  Yes | 11.8 | 0 | 14.3 | 28.6 | 12.9 | 11.1
  No | 88.2 | 100 | 85.7 | 71.4 | 87.1 | 88.9

7. Secondary Outcome: Percentage of Participants With no Increase in BMI SDS at Week 16
Description: Percentage of participants with no increase in BMI SDS at week 16 is presented. In below table, 'Yes' infers percentage of participants with no increase in BMI SDS at week 16 and 'No' infers percentage of participants with increase in BMI SDS at week 16.
Time Frame: At week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 16 | 7 | 34 | 19
Percentage of participants
  Yes | 66.7 | 75.0 | 87.5 | 100 | 76.5 | 84.2
  No | 33.3 | 25.0 | 12.5 | 0 | 23.5 | 15.8

8. Secondary Outcome: Percentage of Participants With no Increase in BMI SDS at Week 52
Description: Percentage of participants with no increase in BMI SDS at week 52 is presented. In below table, 'Yes' infers percentage of participants with no increase in BMI SDS at week 52 and 'No' infers percentage of participants with increase in BMI SDS at week 52.
Time Frame: At week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 14 | 7 | 30 | 16
Percentage of participants
  Yes | 70.6 | 72.7 | 78.6 | 100 | 73.3 | 81.3
  No | 29.4 | 27.3 | 21.4 | 0 | 26.7 | 18.8

9. Secondary Outcome: Change in BMI From Baseline at Week 16
Description: Change in body mass index (BMI) from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram per meter square (kg/m^2)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 16 | 7 | 34 | 19
kilogram per meter square (kg/m^2) | -0.9 (1.4) | -0.8 (1.6) | -1.1 (1.5) | -1.5 (1.7) | -1.0 (1.4) | -1.1 (1.6)

10. Secondary Outcome: Change in BMI From Baseline at Week 52
Description: Change in body mass index (BMI) from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 14 | 7 | 31 | 18
kg/m^2 | 0.8 (2.2) | -0.1 (2.1) | -0.6 (3.3) | -0.7 (2.7) | -0.7 (2.7) | -0.4 (2.3)

11. Secondary Outcome: Change in Body Weight (Kilogram (kg)) From Baseline at Week 16
Description: Change in body weight (kg) from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (kilogram (kg))
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 16 | 7 | 34 | 19
(kilogram (kg)) | -1.7 (3.6) | -1.1 (5.0) | -0.6 (2.2) | -1.0 (2.7) | -1.2 (3.0) | -1.0 (4.2)

12. Secondary Outcome: Change in Body Weight (kg) From Baseline at Week 52
Description: Change in body weight (kg) from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: FAS which included all randomised participants who received at least one dose of trial product and had any post-randomisation data. Overall Number of Participants Analyzed = number of participants who contributed to the analysis. (kilogram (kg))
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 14 | 7 | 31 | 18
kilogram | -0.4 (6.3) | 1.9 (6.0) | 3.0 (6.6) | 2.8 (5.2) | 1.1 (6.5) | 2.3 (5.6)

13. Secondary Outcome: Change in Body Weight (Pounds (lb)) From Baseline at Week 16
Description: Change in body weight (lb) from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pounds (lb)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 16 | 7 | 34 | 19
pounds (lb) | -3.7 (7.8) | -2.4 (11.0) | -1.4 (4.8) | -2.1 (5.9) | -2.6 (6.6) | -2.3 (9.2)

14. Secondary Outcome: Change in Body Weight (lb) From Baseline at Week 52
Description: Change in body weight (lb) from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 14 | 7 | 31 | 18
pounds | -0.9 (13.9) | 4.3 (13.2) | 6.7 (14.4) | 6.2 (11.5) | 2.5 (14.4) | 5.0 (12.3)

15. Secondary Outcome: Change in Body Weight (Percentage [%]) From Baseline at Week 16
Description: Change in body weight (%) from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change in body weight
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 16 | 7 | 34 | 19
Percent change in body weight | -1.7 (3.8) | -0.7 (3.7) | -1.1 (4.1) | -2.2 (5.5) | -1.4 (3.9) | -1.2 (4.3)

16. Secondary Outcome: Change in Body Weight (%) From Baseline at Week 52
Description: Change in body weight (%) from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change in body weight
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 14 | 7 | 31 | 18
Percent change in body weight | -0.4 (6.5) | 2.3 (5.7) | 6.3 (12.1) | 4.9 (8.6) | 2.6 (9.9) | 3.3 (6.9)

17. Secondary Outcome: Change in Waist Circumference From Baseline at Week 16
Description: Change in waist circumference from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 15 | 7 | 33 | 19
centimeters (cm) | -2.50 (4.52) | -2.44 (7.84) | -0.73 (6.14) | -1.04 (4.53) | -1.70 (5.31) | -1.92 (6.70)

18. Secondary Outcome: Change in Waist Circumference From Baseline at Week 52
Description: Change in waist circumference from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 13 | 5 | 30 | 16
centimeter | -2.98 (8.68) | -3.48 (7.32) | 0.45 (8.05) | 0.97 (5.99) | -1.49 (8.45) | -2.09 (7.06)

19. Secondary Outcome: Change in Waist-to-hip Circumference Ratio From Baseline at Week 16
Description: Change in waist-to-hip circumference ratio from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Waist-to-hip circumference ratio
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 15 | 7 | 33 | 19
Waist-to-hip circumference ratio | -0.01 (0.04) | -0.02 (0.06) | 0.00 (0.06) | 0.01 (0.04) | -0.01 (0.05) | -0.01 (0.05)

20. Secondary Outcome: Change in Waist-to-hip Circumference Ratio From Baseline at Week 52
Description: Change in waist-to-hip circumference ratio from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: waist-to-hip circumference ratio
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 13 | 5 | 30 | 16
waist-to-hip circumference ratio | -0.01 (0.06) | -0.04 (0.06) | -0.02 (0.05) | -0.01 (0.07) | -0.02 (0.06) | -0.03 (0.06)

21. Secondary Outcome: Change in Hyperphagia Score: Total Score and Hyperphagic Behaviour, Drive and Severity Score From Baseline at Week 16
Description: Change in hyperphagia score (hyperphagia total score and hyperphagic behaviour, drive and severity score respectively), from baseline to week 16 is presented. The Hyperphagia Questionnaire (HQ)- Total Score. It contains 11 questions which are categorised into 3 subscales; Hyperphagic Behaviour, Hyperphagic Drive, and Hyperphagia Severity. The subscales are summed together to compute the Total Score. The Total Score ranges from 11-55, with higher scores indicating more hyperphagia and a worse outcome. The HQ-Behaviour Factor Score ranges from 5-25, with higher scores indicating more hyperphagic behaviours and a worse outcome. The HQ- Drive Factor Score ranges from 4-20, with higher scores indicating higher hyperphagic drive and a worse outcome. The HQ- Severity Factor Score ranges from 2-10, with higher scores indicating higher severity.
Time Frame: Week 0, week 16
Population: FAS which included all randomised participants who received at least one dose of trial product and had any post-randomisation data. Overall Number of Participants Analyzed = number of participants who contributed to the analysis. Number Analyzed = number of participants with available data. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 19 | 12 | 17 | 7 | 36 | 19
Score on a scale
  Hyperphagia behaviour score: number analyzed (Participants) | 19 | 12 | 15 | 7 | 33 | 19
  Hyperphagia behaviour score | -0.8 (2.01) | -1.7 (4.14) | -1.2 (3.83) | -2.6 (2.07) | -1.0 (2.97) | -2.0 (3.48)
  Hyperphagia drive score: number analyzed (Participants) | 19 | 12 | 13 | 5 | 30 | 16
  Hyperphagia drive score | -0.9 (2.80) | -0.9 (2.61) | -1.8 (2.97) | -2.0 (2.89) | -1.3 (2.87) | -1.3 (2.69)
  Hyperphagia severity score | -0.6 (1.54) | -0.3 (2.46) | -0.1 (1.65) | 0.1 (1.46) | -0.4 (1.59) | -0.2 (2.12)
  Hyperphagia total score | -2.4 (5.55) | -2.9 (5.79) | -3.1 (7.28) | -4.4 (5.65) | -2.7 (6.34) | -3.5 (5.63)

22. Secondary Outcome: Change in Hyperphagia Score: Total Score and Hyperphagic Behaviour, Drive and Severity Score From Baseline at Week 52
Description: Change in hyperphagia score (hyperphagia total score and hyperphagic behaviour, drive and severity score respectively), from baseline to week 52 is presented.The Hyperphagia Questionnaire (HQ)- Total Score. It contains 11 questions which are categorised into 3 subscales; Hyperphagic Behaviour, Hyperphagic Drive, and Hyperphagia Severity. The subscales are summed together to compute the Total Score. The Total Score ranges from 11-55, with higher scores indicating more hyperphagia and a worse outcome. The HQ-Behaviour Factor Score ranges from 5-25, with higher scores indicating more hyperphagic behaviours and a worse outcome. The HQ- Drive Factor Score ranges from 4-20, with higher scores indicating higher hyperphagic drive and a worse outcome. The HQ- Severity Factor Score ranges from 2-10, with higher scores indicating higher severity.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 11 | 14 | 5 | 32 | 16
Score on a scale
  Hyperphagia behaviour score | -0.9 (3.20) | -0.6 (2.62) | -0.7 (4.63) | -2.6 (3.65) | -0.8 (3.82) | -1.3 (3.00)
  Hyperphagia drive score | -2.2 (2.90) | -0.5 (2.42) | -1.1 (3.99) | -1.4 (4.45) | -1.7 (3.41) | -0.8 (3.06)
  Hyperphagia severity score | -1.3 (1.81) | -0.9 (2.51) | -0.4 (2.73) | -1.4 (1.82) | -0.9 (2.27) | -1.1 (2.26)
  Hyperphagia total score | -4.4 (6.57) | -2.1 (6.11) | -2.1 (10.11) | -5.4 (8.32) | -3.4 (8.23) | -3.1 (6.77)

23. Secondary Outcome: Change in High Sensitivity C Reactive Protein (hsCRP) From Baseline at Week 16
Description: Change in hsCRP from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligram per liter (mg/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 11 | 6 | 28 | 18
Milligram per liter (mg/L) | 0.79 (2.58) | -0.57 (6.61) | -2.79 (8.03) | 1.87 (2.12) | -0.61 (5.57) | 0.24 (5.57)

24. Secondary Outcome: Change in High Sensitivity C Reactive Protein (hsCRP) From Baseline at Week 52
Description: Change in hsCRP from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 12 | 5 | 28 | 15
mg/L | 0.25 (2.55) | 0.14 (3.67) | -2.42 (9.19) | -0.37 (0.84) | -0.89 (6.31) | -0.03 (2.99)

25. Secondary Outcome: Change in Total Cholesterol From Baseline at Week 16
Description: Change in Total cholesterol (measured as millimoles per liter (mmol/L) from baseline to week 16 is presented as ratio to baseline.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of total cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 12 | 5 | 29 | 17
Ratio of total cholesterol | 0.99 (0.10) | 1.06 (0.14) | 1.02 (0.11) | 0.97 (0.10) | 1.00 (0.10) | 1.03 (0.14)

26. Secondary Outcome: Change in Total Cholesterol From Baseline at Week 52
Description: Change in total cholesterol (measured as millimoles per liter (mmol/L) from baseline to week 52 is presented as ratio to baseline.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of total cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 12 | 5 | 28 | 15
Ratio of total cholesterol | 1.00 (0.18) | 1.06 (0.15) | 1.01 (0.12) | 1.07 (0.07) | 1.01 (0.15) | 1.06 (0.13)

27. Secondary Outcome: Change in Low Density Lipoprotein (LDL)-Cholesterol From Baseline at Week 16
Description: Change in LDL-cholesterol (measured as mmol/L) from baseline to week 16 is presented as ratio to baseline.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of LDL-cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
Ratio of LDL-cholesterol | 1.01 (0.15) | 1.13 (0.19) | 1.04 (0.17) | 0.96 (0.14) | 1.02 (0.16) | 1.07 (0.19)

28. Secondary Outcome: Change in Low Density Lipoprotein (LDL)-Cholesterol From Baseline at Week 52
Description: Change in LDL-cholesterol (measured as mmol/L) from baseline to week 52 is presented as ratio to baseline.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of LDL-cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 12 | 5 | 28 | 15
Ratio of LDL-cholesterol | 1.02 (0.22) | 1.12 (0.23) | 0.99 (0.19) | 1.06 (0.10) | 1.01 (0.20) | 1.10 (0.19)

29. Secondary Outcome: Change in High Density Lipoprotein (HDL)-Cholesterol From Baseline at Week 16
Description: Change in HDL-cholesterol (measured as mmol/L) from baseline to week 16 is presented as ratio to baseline.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of HDL-cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
Ratio of HDL-cholesterol | 0.96 (0.14) | 1.00 (0.20) | 1.01 (0.14) | 1.12 (0.13) | 0.98 (0.14) | 1.04 (0.19)

30. Secondary Outcome: Change in High Density Lipoprotein (HDL)-Cholesterol From Baseline at Week 52
Description: Change in HDL-cholesterol (measured as mmol/L) from baseline to week 52 is presented as ratio to baseline.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of HDL-cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 12 | 5 | 28 | 15
Ratio of HDL-cholesterol | 0.99 (0.19) | 1.02 (0.17) | 1.06 (0.16) | 1.08 (0.12) | 1.02 (0.18) | 1.04 (0.15)

31. Secondary Outcome: Change in Non-high Density Lipoprotein (Non-HDL) Cholesterol From Baseline at Week 16
Description: Change in non-HDL cholesterol (measured as mmol/L) from baseline to week 16 is presented as ratio to baseline.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of non-HDL cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
Ratio of non-HDL cholesterol | 1.02 (0.16) | 1.09 (0.15) | 1.03 (0.16) | 0.93 (0.12) | 1.02 (0.15) | 1.04 (0.16)

32. Secondary Outcome: Change in Non-high Density Lipoprotein (Non-HDL) Cholesterol From Baseline at Week 52
Description: Change in non-HDL cholesterol (measured as mmol/L) from baseline to week 52 is presented as ratio to baseline.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of non-HDL cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 12 | 5 | 28 | 15
Ratio of non-HDL cholesterol | 1.02 (0.22) | 1.07 (0.19) | 1.00 (0.16) | 1.07 (0.13) | 1.01 (0.19) | 1.07 (0.17)

33. Secondary Outcome: Change in Very Low-density Lipoprotein (VLDL) Cholesterol From Baseline at Week 16
Description: Change in VLDL cholesterol (measured as mmol/L) from baseline to week 16 is presented as ratio to baseline.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of VLDL cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 12 | 5 | 29 | 17
Ratio of VLDL cholesterol | 1.05 (0.36) | 0.98 (0.27) | 1.05 (0.46) | 0.80 (0.17) | 1.05 (0.40) | 0.93 (0.25)

34. Secondary Outcome: Change in Very Low-density Lipoprotein (VLDL) Cholesterol From Baseline at Week 52
Description: Change in VLDL cholesterol (measured as mmol/L) from baseline to week 52 is presented as ratio to baseline.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of VLDL cholesterol
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 12 | 5 | 28 | 15
Ratio of VLDL cholesterol | 1.06 (0.35) | 0.95 (0.36) | 1.03 (0.26) | 1.13 (0.31) | 1.04 (0.31) | 1.01 (0.34)

35. Secondary Outcome: Change in Triglycerides From Baseline at Week 16
Description: Change in triglycerides (measured as mmol/L) from baseline to week 16 is presented as ratio to baseline.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of triglycerides
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 12 | 5 | 29 | 17
Ratio of triglycerides | 1.04 (0.36) | 0.99 (0.26) | 1.05 (0.44) | 0.80 (0.18) | 1.05 (0.39) | 0.93 (0.25)

36. Secondary Outcome: Change in Triglycerides From Baseline at Week 52
Description: Change in triglycerides (measured as mmol/L) from baseline to week 52 is presented as ratio to baseline.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of triglycerides
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 12 | 5 | 28 | 15
Ratio of triglycerides | 1.07 (0.36) | 0.94 (0.36) | 1.04 (0.29) | 1.12 (0.32) | 1.06 (0.32) | 1.00 (0.35)

37. Secondary Outcome: Change in Fasting Lipid: Free Fatty Acids (FFA) From Baseline at Week 16
Description: Change in free fatty acids (measured as mmol/L) from baseline to week 16 is presented as ratio to baseline.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of FFA
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 11 | 13 | 5 | 29 | 16
Ratio of FFA | 1.52 (1.60) | 1.31 (0.61) | 1.04 (0.35) | 0.99 (0.30) | 1.31 (1.21) | 1.21 (0.55)

38. Secondary Outcome: Change in Fasting Lipid: Free Fatty Acids (FFA) From Baseline at Week 52
Description: Change in free fatty acids (measured as mmol/L) from baseline to week 52 is presented as ratio to baseline.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of FFA
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 15 | 8 | 12 | 4 | 27 | 12
Ratio of FFA | 1.15 (0.76) | 1.45 (0.49) | 0.85 (0.51) | 1.05 (0.25) | 1.01 (0.67) | 1.32 (0.45)

39. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure From Baseline at Week 16
Description: Change in systolic blood pressure (SBP) and diastolic blood pressure (DBP) from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 15 | 7 | 33 | 19
Millimeters of mercury (mmHg)
  SBP: Change from week 0 to week 16 | -5 (15) | -2 (13) | 2 (9) | 2 (6) | -1 (13) | -1 (11)
  DBP: Change from week 0 to week 16 | -1 (10) | 0 (7) | 1 (8) | -1 (17) | 0 (9) | 0 (11)

40. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure From Baseline at Week 52
Description: Change in systolic blood pressure (SBP) and diastolic blood pressure (DBP) from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 13 | 5 | 30 | 16
Millimeters of mercury (mmHg)
  SBP: Change from week 0 to week 52 | -5 (6) | 4 (12) | 4 (15) | 7 (8) | -1 (11) | 5 (11)
  DBP: Change from week 0 to week 52 | -3 (9) | 5 (13) | 4 (13) | 1 (7) | 0 (11) | 4 (12)

41. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline at Week 16
Description: Change in HbA1c from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 12 | 13 | 7 | 29 | 19
Percentage point of HbA1c | -0.2 (0.1) | 0 (0.3) | -0.2 (0.3) | -0.2 (0.3) | -0.2 (0.2) | -0.1 (0.3)

42. Secondary Outcome: Change in HbA1c From Baseline at Week 52
Description: Change in HbA1c from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 9 | 12 | 5 | 28 | 14
Percentage point of HbA1c | -0.2 (0.2) | 0.1 (0.3) | -0.2 (0.4) | -0.1 (0.3) | -0.2 (0.3) | 0.1 (0.3)

43. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline at Week 16
Description: Change in FPG from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 11 | 13 | 5 | 31 | 16
mmol/L | -0.2 (0.5) | 0.1 (0.5) | -0.1 (0.5) | 0.2 (0.4) | -0.2 (0.5) | 0.1 (0.4)

44. Secondary Outcome: Change in FPG From Baseline at Week 52
Description: Change in FPG from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 15 | 9 | 12 | 5 | 27 | 14
mmol/L | 0 (0.7) | 0.3 (0.8) | 0 (0.4) | 0 (0.4) | 0 (0.6) | 0.2 (0.7)

45. Secondary Outcome: Change in Fasting Insulin From Baseline at Week 16
Description: Change in fasting insulin (measured as picomoles per litre (pmol/L)) from baseline to week 16 is presented as ratio to baseline.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of fasting insulin
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 11 | 13 | 6 | 31 | 17
Ratio of fasting insulin | 1.59 (1.91) | 0.78 (0.32) | 1.43 (1.17) | 1.32 (0.68) | 1.52 (1.62) | 0.97 (0.53)

46. Secondary Outcome: Change in Fasting Insulin From Baseline at Week 52
Description: Change in fasting insulin (measured as picomoles per litre (pmol/L)) from baseline to week 52 is presented as ratio to baseline.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of fasting insulin
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 8 | 12 | 5 | 28 | 13
Ratio of fasting insulin | 2.03 (2.33) | 0.79 (0.37) | 1.45 (1.27) | 1.22 (0.44) | 1.78 (1.94) | 0.96 (0.44)

47. Secondary Outcome: Change in Fasting C Peptide From Baseline at Week 16
Description: Change in fasting C peptide (measured as nano moles per liter (nmol/L)) from baseline to week 16 is presented as ratio to baseline.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of fasting C peptide
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 11 | 12 | 6 | 30 | 17
Ratio of fasting C peptide | 1.14 (0.56) | 0.86 (0.20) | 1.11 (0.50) | 1.08 (0.44) | 1.13 (0.53) | 0.94 (0.31)

48. Secondary Outcome: Change in Fasting C Peptide From Baseline at Week 52
Description: Change in fasting C peptide (measured as nano moles per liter (nmol/L)) from baseline to week 52 is presented as ratio to baseline.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of fasting C peptide
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 8 | 12 | 5 | 28 | 13
Ratio of fasting C peptide | 1.34 (0.92) | 0.91 (0.23) | 1.15 (0.45) | 1.09 (0.30) | 1.26 (0.75) | 0.98 (0.26)

49. Secondary Outcome: Number of Participants in Glycaemic Category at Week 16
Description: Number of participants in glycaemic categories, "normoglycaemia, pre-diabetes and type 2 diabetes" at Week 16 are presented. These categories were set as per the following criteria: 1) Normoglycaemia: FPG <5.6 mmol/L (<100 mg/dL) and/or HbA1c <5.7%. 2) Pre-diabetes: FPG 5.6-6.9 mmol/L (both inclusive), FPG 100-125 mg/dL (both inclusive) or HbA1c 5.7-6.4% (both inclusive). 3) Type 2 diabetes: FPG ≥7.0 mmol/L (≥126 mg/dL) and/or HbA1c ≥6.5%.
Time Frame: week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 13 | 7 | 31 | 19
Participants
  Normoglycaemia | 16 | 8 | 11 | 5 | 27 | 13
  Pre-diabetes | 2 | 4 | 2 | 2 | 4 | 6
  Type 2 diabetes | 0 | 0 | 0 | 0 | 0 | 0

50. Secondary Outcome: Number of Participants in Glycaemic Category at Week 52
Description: Number of participants in glycaemic categories, "normoglycaemia, pre-diabetes and type 2 diabetes" at Week 52 are presented. These categories were set as per the following criteria: 1) Normoglycaemia: FPG <5.6 mmol/L (<100 mg/dL) and/or HbA1c <5.7%. 2) Pre-diabetes: FPG 5.6-6.9 mmol/L (both inclusive), FPG 100-125 mg/dL (both inclusive) or HbA1c 5.7-6.4% (both inclusive). 3) Type 2 diabetes: FPG ≥7.0 mmol/L (≥126 mg/dL) and/or HbA1c ≥6.5%.
Time Frame: Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 9 | 12 | 5 | 28 | 14
Participants
  Normoglycaemia | 13 | 4 | 10 | 2 | 23 | 6
  Pre-diabetes | 2 | 4 | 2 | 3 | 4 | 7
  Type 2 diabetes | 1 | 1 | 0 | 0 | 1 | 1

51. Secondary Outcome: Change in Homeostasis Model Assessment of Beta-cell Function (HOMA-B) From Baseline at Week 16
Description: Change in HOMA-B from baseline to week 16 is presented as ratio to baseline. HOMA-B was calculated as: Beta-cell function (%) = 20·fasting insulin[mU/L]/(FPG[mmol/L]-3.5).
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of HOMA-B
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 10 | 13 | 5 | 31 | 15
Ratio of HOMA-B | 1.69 (1.93) | 0.70 (0.31) | 1.55 (1.04) | 1.07 (0.51) | 1.63 (1.59) | 0.82 (0.41)

52. Secondary Outcome: Change in Homeostasis Model Assessment of Beta-cell Function (HOMA-B) From Baseline at Week 52
Description: Change in HOMA-B from baseline to week 52 is presented as ratio to baseline. HOMA-B was calculated as: Beta-cell function (%) = 20·fasting insulin[mU/L]/(FPG[mmol/L]-3.5).
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of HOMA-B
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 15 | 8 | 12 | 5 | 27 | 13
Ratio of HOMA-B | 2.24 (1.85) | 0.65 (0.30) | 1.50 (1.50) | 1.25 (0.50) | 1.91 (1.71) | 0.88 (0.48)

53. Secondary Outcome: Change in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) From Baseline at Week 16
Description: Change in HOMA-IR from baseline to week 16 is presented as ratio to baseline. HOMA-IR was calculated as: Insulin resistance (%) = fasting plasma glucose [mmol/L] x fasting insulin [mmol/L]/ 22.5.
Time Frame: Week 0, week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of HOMA-IR
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 10 | 13 | 5 | 31 | 15
Ratio of HOMA-IR | 1.57 (1.92) | 0.80 (0.35) | 1.43 (1.26) | 1.33 (0.82) | 1.51 (1.65) | 0.97 (0.58)

54. Secondary Outcome: Change in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) From Baseline at Week 52
Description: Change in HOMA-IR from baseline to week 52 is presented as ratio to baseline. HOMA-IR was calculated as: Insulin resistance (%) = fasting plasma glucose [mmol/L] x fasting insulin [mmol/L]/ 22.5.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of HOMA-IR
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 15 | 8 | 12 | 5 | 27 | 13
Ratio of HOMA-IR | 2.26 (3.13) | 0.88 (0.50) | 1.45 (1.23) | 1.24 (0.48) | 1.90 (2.46) | 1.02 (0.51)

55. Secondary Outcome: Number of Treatment Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial participant administered or using a medicinal product, whether or not considered related to the medicinal product or usage. All AEs reported here are TEAEs. TEAE is defined as an event that had onset date during the on-treatment period. The endpoint was evaluated based on the data from on-treatment period. On-treatment period included AEs are with an onset date on or after the first day of trial product administration and any of the following dates, whichever came first: a) 14 days after the last day on trial product, or b) Follow-up visit (week 54) for participants with trial product discontinuation, or c) Last study visit (participants withdrawn without follow-up visit (week 54)).
Time Frame: From week 0 to week 54
Population: Safety analysis set (SAS) which included all participants exposed to at least one dose of trial product. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Number; unit: Events
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 20 | 12 | 17 | 7 | 37 | 19
Events | 134 | 37 | 159 | 8 | 293 | 45

56. Secondary Outcome: Number of Severe Treatment Emergent Episodes of Hypoglycaemia
Description: Hypoglycaemic episode (blood glucose less than or equal to (<=) 3.9 mmol/L (70 mg/dL) Or greater than (>) 3.9 mmol/L (70 mg/dL) occurring in conjunction with hypoglycaemic symptoms) is defined as treatment emergent if the onset of the episode was on or after the first day of exposure to randomised treatment and no later than 14 days after the last day on randomised treatment. Severe hypoglycaemia defined by American Diabetes Association (ADA) 2013 and International Society for Paediatric and Adolescent Diabetes (ISPAD) 2018: hypoglycaemic episode associated with severe cognitive impairment requiring external assistance for recovery. Endpoint was evaluated based on data from in-trial period which was defined as events with onset date on or after the first day of trial product administration and no later than the last study visit (week 54).
Time Frame: From week 0 to week 54
Population: SAS which included all participants exposed to at least one dose of trial product. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Number; unit: Episodes
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 20 | 12 | 17 | 7 | 37 | 19
Episodes | 0 | 0 | 1 | 0 | 1 | 0

57. Secondary Outcome: Number of Blood Glucose Confirmed Symptomatic Episodes of Hypoglycaemia
Description: Symptomatic blood glucose confirmed hypoglycaemia: An episode that is blood glucose confirmed by plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Hypoglycaemic episode is defined as treatment emergent if the onset of the episode was on or after the first day of exposure to randomised treatment and no later than 14 days after the last day on randomised treatment. Endpoint was evaluated based on data from in-trial period which was defined as events with onset date on or after the first day of trial product administration and no later than the last study visit (week 54).
Time Frame: From week 0 to week 54
Population: as for outcome 56
Measure: Number; unit: Episodes
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 20 | 12 | 17 | 7 | 37 | 19
Episodes | 0 | 0 | 0 | 0 | 0 | 0

58. Secondary Outcome: Number of Participants With Occurrence of Anti-liraglutide Antibodies
Description: Number of participants with occurrence of anti-liraglutide antibodies is presented. In the below table, 'Yes' infers number of participants with occurrence of anti- liraglutide antibodies and 'No' infers number of participants without anti- liraglutide antibodies.
Time Frame: From week 0 to week 54
Population: SAS which included all participants exposed to at least one dose of trial product. Overall number of participants analysed = Number of participants with available data. Combined data of Part A and B for liraglutide was planned to be reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part B: Liraglutide | Part A+B: Liraglutide
Number analyzed (Participants) | 16 | 9 | 25
Participants
  Yes | 2 | 1 | 3
  No | 14 | 8 | 22

59. Secondary Outcome: Number of Participants With Change in Electrocardiogram (ECG) From Baseline at Week 16
Description: A 12-lead ECG was performed at baseline (week 0) and week 16 and categorised as normal, abnormal and not clinically significant (abnormal NCS) or abnormal and clinically significant (abnormal CS). Number of participants in each ECG category at week 0 and weeks 16 are presented.
Time Frame: Week 0, Week 16
Population: SAS which included all participants exposed to at least one dose of trial product. Number Analyzed = number of participants with available data. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 20 | 12 | 17 | 7 | 37 | 19
Participants
  Week 0: Normal | 20 | 12 | 17 | 6 | 37 | 18
  Week 0: Abnormal, NCS | 0 | 0 | 0 | 1 | 0 | 1
  Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: Normal: number analyzed (Participants) | 17 | 12 | 14 | 7 | 31 | 19
  Week 16: Normal | 17 | 12 | 13 | 7 | 30 | 19
  Week 16: Abnormal, NCS: number analyzed (Participants) | 17 | 12 | 14 | 7 | 31 | 19
  Week 16: Abnormal, NCS | 0 | 0 | 1 | 0 | 1 | 0
  Week 16: Abnormal, CS: number analyzed (Participants) | 17 | 12 | 14 | 7 | 31 | 19
  Week 16: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0

60. Secondary Outcome: Number of Participants With Change in ECG From Baseline at Week 52
Description: A 12-lead ECG was performed at baseline (week 0) and week 52 and categorised as normal, abnormal and not clinically significant (abnormal NCS) or abnormal and clinically significant (abnormal CS). Number of participants in each ECG category at week 0 and week 52 are presented.
Time Frame: Week 0, Week 52
Population: as for outcome 59
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 20 | 12 | 17 | 7 | 37 | 19
Participants
  Week 0: Normal | 20 | 12 | 17 | 6 | 37 | 18
  Week 0: Abnormal, NCS | 0 | 0 | 0 | 1 | 0 | 1
  Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Week 52: Normal: number analyzed (Participants) | 18 | 10 | 13 | 4 | 31 | 14
  Week 52: Normal | 17 | 9 | 13 | 4 | 30 | 13
  Week 52: Abnormal, NCS: number analyzed (Participants) | 18 | 10 | 13 | 4 | 31 | 14
  Week 52: Abnormal, NCS | 1 | 1 | 0 | 0 | 1 | 1
  Week 52: Abnormal, CS: number analyzed (Participants) | 18 | 10 | 13 | 4 | 31 | 14
  Week 52: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0

61. Secondary Outcome: Change in Pulse From Baseline at Week 16
Description: Change in pulse from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: SAS which included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = number of participants with available data. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 15 | 7 | 33 | 19
Beats/minute | 2 (12) | -2 (5) | 1 (16) | -9 (10) | 2 (14) | -4 (8)

62. Secondary Outcome: Change in Pulse From Baseline at Week 52
Description: Change in pulse from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 13 | 5 | 30 | 16
Beats/minute | 1 (13) | -8 (10) | 10 (11) | -6 (8) | 5 (13) | -7 (10)

63. Secondary Outcome: Change in Haematology: Haemoglobin From Baseline at Week 16
Description: Change in haemoglobin from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 11 | 12 | 6 | 28 | 17
millimoles per liter (mmol/L) | -0.18 (0.43) | 0.06 (0.28) | -0.20 (1.22) | -0.07 (0.55) | -0.19 (0.84) | 0.01 (0.38)

64. Secondary Outcome: Change in Haematology: Haemoglobin From Baseline at Week 52
Description: Change in haemoglobin from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 15 | 9 | 10 | 4 | 25 | 13
mmol/L | -0.14 (0.79) | -0.01 (0.31) | -0.02 (0.61) | -0.02 (0.20) | -0.09 (0.72) | -0.01 (0.28)

65. Secondary Outcome: Change in Haematology: Haematocrit From Baseline at Week 16
Description: Change in haematocrit from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: Percentage of haematocrit in blood
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 11 | 12 | 6 | 28 | 17
Percentage of haematocrit in blood | -1.8 (2.1) | -0.5 (1.3) | 0.4 (2.6) | -0.6 (3.3) | -0.9 (2.6) | -0.5 (2.1)

66. Secondary Outcome: Change in Haematology: Haematocrit From Baseline at Week 52
Description: Change in haematocrit from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: Percentage of haematocrit in blood
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 15 | 9 | 10 | 4 | 25 | 13
Percentage of haematocrit in blood | -1.4 (4.0) | 0 (1.7) | -0.2 (2.7) | -0.8 (2.6) | -0.9 (3.5) | -0.3 (1.9)

67. Secondary Outcome: Change in Haematology: Thrombocytes, Leukocytes, Eosinophils, Neutrophils, Basophils, Lymphocytes, Monocytes From Baseline at Week 16
Description: Change in thrombocytes, leukocytes, eosinophils, neutrophils, basophils, lymphocytes, monocytes from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: SAS which included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = number of participants who contributed to the analysis. Number Analyzed = number of participants with available data. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 11 | 12 | 6 | 28 | 17
10^9 cells per liter (10^9/L)
  Thrombocytes: Change from week 0 to week 16: number analyzed (Participants) | 16 | 11 | 11 | 5 | 27 | 16
  Thrombocytes: Change from week 0 to week 16 | 6 (35) | -21 (26) | 8 (66) | 19 (18) | 7 (49) | -8 (30)
  Leukocytes: Change from week 0 to week 16 | -0.1 (1.5) | -0.3 (1.6) | -0.8 (2.3) | -1.1 (1.7) | -0.4 (1.9) | -0.6 (1.6)
  Eosinophils: Change from week 0 to week 16 | -0.03 (0.09) | 0.04 (0.07) | -0.14 (0.27) | 0.07 (0.32) | -0.07 (0.20) | 0.05 (0.19)
  Neutrophils: Change from week 0 to week 16 | 0.11 (1.08) | -0.22 (1.62) | -0.28 (1.59) | -1.35 (1.33) | -0.06 (1.31) | -0.62 (1.58)
  Basophils: Change from week 0 to week 16 | -0.01 (0.02) | 0 (0.02) | -0.01 (0.04) | -0.01 (0.04) | -0.01 (0.03) | 0 (0.03)
  Lymphocytes: Change from week 0 to week 16 | -0.24 (0.66) | -0.09 (0.97) | -0.36 (0.89) | 0.09 (0.85) | -0.29 (0.76) | -0.02 (0.91)
  Monocytes: Change from week 0 to week 16 | 0.06 (0.17) | -0.04 (0.12) | -0.05 (0.17) | 0.05 (0.20) | 0.01 (0.18) | -0.01 (0.15)

68. Secondary Outcome: Change in Haematology: Thrombocytes, Leukocytes, Eosinophils, Neutrophils, Basophils, Lymphocytes, Monocytes From Baseline at Week 52
Description: Change in thrombocytes, leukocytes, eosinophils, neutrophils, basophils, lymphocytes, monocytes from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 15 | 9 | 10 | 4 | 25 | 13
10^9 cells per liter (10^9/L)
  Thrombocytes: Change from week 0 to week 52: number analyzed (Participants) | 15 | 8 | 9 | 3 | 24 | 11
  Thrombocytes: Change from week 0 to week 52 | 18 (44) | -7 (39) | -2 (37) | 37 (70) | 10 (42) | 5 (49)
  Leukocytes: Change from week 0 to week 52 | -0.2 (1.1) | -0.6 (1.7) | -0.7 (2.8) | 0.3 (3.0) | -0.4 (1.9) | -0.3 (2.1)
  Eosinophils: Change from week 0 to week 52 | 0.01 (0.11) | 0.03 (0.19) | -0.13 (0.36) | -0.17 (0.13) | -0.05 (0.24) | -0.03 (0.20)
  Neutrophils: Change from week 0 to week 52 | 0.11 (1.17) | -0.76 (1.40) | -0.03 (2.03) | -0.07 (2.55) | 0.05 (1.53) | -0.55 (1.75)
  Basophils: Change from week 0 to week 52 | 0 (0.03) | 0 (0.04) | -0.01 (0.04) | 0.02 (0.04) | -0.01 (0.04) | 0.01 (0.04)
  Lymphocytes: Change from week 0 to week 52 | -0.28 (0.67) | 0.19 (0.70) | -0.47 (0.59) | 0.39 (0.49) | -0.36 (0.63) | 0.25 (0.63)
  Monocytes: Change from week 0 to week 52 | -0.04 (0.19) | -0.06 (0.22) | -0.05 (0.19) | 0.14 (0.20) | -0.04 (0.19) | 0 (0.23)

69. Secondary Outcome: Change in Haematology: Erythrocytes From Baseline at Week 16
Description: Change in erythrocytes from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: SAS which included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = number of participants who contributed to the analysis. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 11 | 12 | 6 | 28 | 17
10^12 cells per liter (10^12/L) | -0.1 (0.2) | 0 (0.2) | 0.1 (0.3) | 0 (0.3) | -0.1 (0.3) | 0 (0.2)

70. Secondary Outcome: Change in Haematology: Erythrocytes From Baseline at Week 52
Description: Change in erythrocytes from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 15 | 9 | 10 | 4 | 25 | 13
10^12 cells per liter (10^12/L) | -0.1 (0.4) | 0 (0.2) | -0.1 (0.3) | 0 (0) | -0.1 (0.4) | 0 (0.1)

71. Secondary Outcome: Change in Biochemistry: Creatinine and Bilirubin (Total) From Baseline at Week 16
Description: Change in creatinine and bilirubin (total) from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: micro mole per liter (umol/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 11 | 6 | 28 | 18
micro mole per liter (umol/L)
  Creatinine: Change from week 0 to week 16: number analyzed (Participants) | 17 | 12 | 10 | 6 | 27 | 18
  Creatinine: Change from week 0 to week 16 | 1 (5) | 0 (6) | 2 (7) | 0 (6) | 1 (5) | 0 (6)
  Bilirubin (total): Change from week 0 to week 16: number analyzed (Participants) | 17 | 12 | 11 | 5 | 28 | 17
  Bilirubin (total): Change from week 0 to week 16 | 0 (2) | 0 (2) | 0 (2) | 1 (2) | 0 (2) | 0 (2)

72. Secondary Outcome: Change in Biochemistry: Creatinine and Bilirubin (Total) From Baseline at Week 52
Description: Change in creatinine and bilirubin (total) from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 11 | 5 | 27 | 15
umol/L
  Creatinine: Change from week 0 to week 52 | 3 (8) | -4 (9) | 3 (6) | 5 (3) | 3 (7) | -1 (9)
  Bilirubin (total): Change from week 0 to week 52 | 0 (2) | 2 (3) | 0 (1) | 2 (3) | 0 (2) | 2 (3)

73. Secondary Outcome: Change in Biochemistry: Creatine Kinase, Amylase, Lipase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP) From Baseline at Week 16
Description: Change in creatine kinase, amylase, lipase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 11 | 6 | 28 | 18
Units per liter (U/L)
  Creatinine kinase: Change from week 0 to week 16: number analyzed (Participants) | 17 | 12 | 11 | 5 | 28 | 17
  Creatinine kinase: Change from week 0 to week 16 | -3 (37) | 16 (45) | 3 (23) | -5 (5) | -1 (32) | 10 (39)
  Amylase: Change from week 0 to week 16 | 5 (13) | -2 (5) | 8 (12) | 8 (8) | 6 (13) | 1 (8)
  Lipase: Change from week 0 to week 16 | 10 (6) | 0 (4) | 8 (7) | 1 (2) | 9 (6) | 0 (3)
  ALT: Change from week 0 to week 16: number analyzed (Participants) | 17 | 12 | 11 | 5 | 28 | 17
  ALT: Change from week 0 to week 16 | -9 (32) | -4 (18) | -2 (6) | -25 (23) | -6 (25) | -10 (21)
  AST: Change from week 0 to week 16: number analyzed (Participants) | 16 | 12 | 11 | 5 | 27 | 17
  AST: Change from week 0 to week 16 | -6 (14) | 0 (10) | -2 (5) | -18 (24) | -4 (11) | -6 (17)
  ALP: Change from week 0 to week 16: number analyzed (Participants) | 17 | 12 | 10 | 5 | 27 | 17
  ALP: Change from week 0 to week 16 | -10 (12) | -7 (25) | -21 (36) | -47 (42) | -14 (24) | -19 (35)

74. Secondary Outcome: Change in Biochemistry: Creatine Kinase, Amylase, Lipase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP) From Baseline at Week 52
Description: Change in creatine kinase, amylase, lipase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 11 | 5 | 27 | 15
Units per liter (U/L)
  Creatinine kinase: Change from week 0 to week 52 | 30 (206) | -4 (29) | 25 (42) | -8 (25) | 28 (159) | -5 (27)
  Amylase: Change from week 0 to week 52 | 4 (10) | 2 (12) | 7 (12) | 8 (5) | 5 (11) | 4 (11)
  Lipase: Change from week 0 to week 52 | 9 (9) | -1 (3) | 7 (6) | 3 (5) | 8 (8) | 0 (4)
  ALT: Change from week 0 to week 52: number analyzed (Participants) | 16 | 9 | 11 | 5 | 27 | 14
  ALT: Change from week 0 to week 52 | 1 (12) | 4 (25) | 0 (16) | -24 (28) | 1 (14) | -6 (29)
  AST: Change from week 0 to week 52: number analyzed (Participants) | 15 | 9 | 11 | 4 | 26 | 13
  AST: Change from week 0 to week 52 | -2 (7) | 9 (31) | 1 (7) | -21 (32) | -1 (7) | 0 (33)
  ALP: Change from week 0 to week 52 | -24 (27) | -35 (27) | -25 (59) | -26 (60) | -24 (42) | -32 (39)

75. Secondary Outcome: Change in Biochemistry: Urea, Sodium, Potassium, Calcium Total and Calcium Albumin-corrected From Baseline at Week 16
Description: Change in urea, sodium, potassium, calcium total and calcium albumin-corrected from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 11 | 6 | 28 | 18
mmol/L
  Urea: Change from week 0 to week 16 | 0.03 (1.45) | -0.51 (0.67) | 0 (0.99) | 0.09 (2.19) | 0.02 (1.26) | -0.31 (1.33)
  Sodium: Change from week 0 to week 16: number analyzed (Participants) | 17 | 12 | 10 | 6 | 27 | 18
  Sodium: Change from week 0 to week 16 | 0 (5) | 2 (3) | 1 (4) | 0 (1) | 0 (4) | 1 (3)
  Potassium: Change from week 0 to week 16: number analyzed (Participants) | 16 | 12 | 10 | 6 | 26 | 18
  Potassium: Change from week 0 to week 16 | 0.1 (0.4) | -0.1 (0.3) | -0.2 (0.6) | -0.1 (0.2) | 0 (0.5) | -0.1 (0.2)
  Calcium: Change from week 0 to week 16 | 0 (0.12) | 0 (0.10) | 0.08 (0.17) | 0.02 (0.10) | 0.03 (0.14) | 0.01 (0.10)

76. Secondary Outcome: Change in Biochemistry: Urea, Sodium, Potassium, Calcium Total and Calcium Albumin-corrected From Baseline at Week 52
Description: Change in urea, sodium, potassium, calcium total and calcium albumin-corrected from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 11 | 5 | 27 | 15
mmol/L
  Urea: Change from week 0 to week 52 | -0.38 (1.56) | -0.34 (0.54) | -0.21 (1.00) | -0.04 (1.08) | -0.31 (1.34) | -0.24 (0.74)
  Sodium: Change from week 0 to week 52 | -1 (5) | -2 (5) | 1 (4) | 2 (2) | 0 (4) | -1 (4)
  Potassium: Change from week 0 to week 52: number analyzed (Participants) | 15 | 9 | 11 | 5 | 26 | 14
  Potassium: Change from week 0 to week 52 | -0.2 (0.6) | -0.1 (0.2) | -0.2 (0.7) | 0 (0.2) | -0.2 (0.6) | -0.1 (0.2)
  Calcium: Change from week 0 to week 52 | -0.05 (0.14) | -0.11 (0.12) | 0.09 (0.14) | 0 (0.02) | 0.01 (0.15) | -0.08 (0.11)

77. Secondary Outcome: Change in Biochemistry: Albumin From Baseline at Week 16
Description: Change in albumin from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 11 | 5 | 28 | 17
gram per deciliter (g/dL) | 0 (0.2) | 0 (0.1) | 0 (0.2) | 0 (0.1) | 0 (0.2) | 0 (0.1)

78. Secondary Outcome: Change in Biochemistry: Albumin From Baseline at Week 52
Description: Change in albumin from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 11 | 5 | 27 | 15
g/dL | -0.1 (0.7) | -0.1 (0.3) | 0 (0.2) | 0 (0.1) | 0 (0.5) | -0.1 (0.2)

79. Secondary Outcome: Change in Hormone Level: Carcinoembryonic Antigen (CEA) From Baseline at Week 16
Description: Change in CEA serum from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 9 | 13 | 6 | 30 | 15
nanogram per milliliter (ng/mL) | -0.01 (0.11) | -0.17 (0.30) | 0.17 (0.55) | -0.04 (0.10) | 0.07 (0.38) | -0.12 (0.24)

80. Secondary Outcome: Change in Hormone Level: Carcinoembryonic Antigen (CEA) From Baseline at Week 52
Description: Change in CEA serum from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 15 | 7 | 12 | 5 | 27 | 12
ng/mL | 0.03 (0.38) | -0.14 (0.26) | -0.01 (0.14) | 0.17 (0.24) | 0.01 (0.29) | -0.01 (0.29)

81. Secondary Outcome: Change in Hormone Level: Calcitonin From Baseline at Week 16
Description: Change in calcitonin from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 11 | 6 | 28 | 17
nanogram per liter (ng/L) | 0 (0) | 0 (0) | 0.3 (1.1) | 0 (0) | 0.1 (0.7) | 0 (0)

82. Secondary Outcome: Change in Hormone Level: Calcitonin From Baseline at Week 52
Description: Change in calcitonin from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 7 | 11 | 5 | 27 | 12
ng/L | 0.1 (0.6) | 0 (0) | 0.5 (1.2) | 0 (0) | 0.3 (0.9) | 0 (0)

83. Secondary Outcome: Change in Hormone Level: Thyroid Stimulating Hormone (TSH) and Prolactin From Baseline at Week 16
Description: Change in TSH and prolactin from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Milli-international units/liter (mIU/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 13 | 7 | 30 | 19
Milli-international units/liter (mIU/L)
  TSH: Change from week 0 to week 16: number analyzed (Participants) | 17 | 12 | 12 | 7 | 29 | 19
  TSH: Change from week 0 to week 16 | -0.34 (0.68) | -0.01 (0.72) | -0.09 (1.13) | -0.59 (0.67) | -0.23 (0.89) | -0.23 (0.74)
  Prolactin: Change from week 0 to week 16 | 7 (27) | -6 (33) | 0 (13) | -22 (63) | 4 (22) | -12 (45)

84. Secondary Outcome: Change in Hormone Level: Thyroid Stimulating Hormone (TSH) and Prolactin From Baseline at Week 52
Description: Change in TSH and prolactin from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 11 | 5 | 27 | 15
mIU/L
  TSH: Change from week 0 to week 52 | 0.02 (1.59) | -0.48 (0.63) | -0.75 (2.13) | -0.17 (1.08) | -0.30 (1.83) | -0.38 (0.78)
  Prolactin: Change from week 0 to week 52 | 10 (38) | 8 (37) | -3 (37) | 29 (33) | 5 (37) | 15 (36)

85. Secondary Outcome: Change in Hormone Level: Free Thyroxine (Free T4) and Adrenocorticotropic Hormone (ACTH) From Baseline at Week 16
Description: Change in free T4 and ACTH from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 13 | 7 | 31 | 19
picomole per liter (pmol/L)
  T4: Change from week 0 to week 16: number analyzed (Participants) | 17 | 12 | 13 | 7 | 30 | 19
  T4: Change from week 0 to week 16 | -0.6 (1.4) | 0.3 (1.1) | 0.7 (2.3) | 0.1 (1.7) | -0.1 (1.9) | 0.2 (1.3)
  ACTH: Change from week 0 to week 16: number analyzed (Participants) | 18 | 9 | 13 | 5 | 31 | 14
  ACTH: Change from week 0 to week 16 | 0.99 (5.22) | -0.85 (2.22) | -0.37 (1.49) | -1.32 (1.87) | 0.42 (4.10) | -1.02 (2.04)

86. Secondary Outcome: Change in Hormone Level: Free Thyroxine (Free T4) and Adrenocorticotropic Hormone (ACTH) From Baseline at Week 52
Description: Change in free T4 and ACTH from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 12 | 5 | 27 | 15
pmol/L
  T4: Change from week 0 to week 52: number analyzed (Participants) | 16 | 10 | 11 | 5 | 27 | 15
  T4: Change from week 0 to week 52 | -0.4 (1.7) | 1.9 (2.7) | -0.1 (2.0) | 0.8 (2.3) | -0.3 (1.8) | 1.5 (2.5)
  ACTH: Change from week 0 to week 52: number analyzed (Participants) | 15 | 7 | 12 | 4 | 27 | 11
  ACTH: Change from week 0 to week 52 | -0.02 (2.02) | 1.29 (3.50) | 0.98 (5.64) | 0.20 (2.41) | 0.42 (3.99) | 0.89 (3.07)

87. Secondary Outcome: Change in Hormone Level: Insulin-like Growth Factor-1 (IGF-1) and Cortisol From Baseline at Week 16
Description: Change in IGF-1 and cortisol from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 11 | 13 | 7 | 31 | 18
nanogram per milliliter (ng/mL)
  IGF-1: Change from week 0 to week 16: number analyzed (Participants) | 16 | 11 | 13 | 5 | 29 | 16
  IGF-1: Change from week 0 to week 16 | -56.89 (126.46) | -28.23 (95.79) | 2.41 (84.98) | -14.23 (75.01) | -30.31 (112.09) | -23.86 (87.54)
  Cortisol: Change from week 0 to week 16 | -22.94 (41.36) | 6.75 (38.72) | -8.09 (22.98) | -23.08 (59.02) | -16.71 (35.16) | -4.85 (48.33)

88. Secondary Outcome: Change in Hormone Level: Insulin-like Growth Factor-1 (IGF-1) and Cortisol From Baseline at Week 52
Description: Change in IGF-1 and cortisol from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 9 | 12 | 5 | 28 | 14
ng/mL
  IGF-1: Change from week 0 to week 52: number analyzed (Participants) | 15 | 8 | 12 | 5 | 27 | 13
  IGF-1: Change from week 0 to week 52 | -25.90 (195.61) | -103.45 (136.61) | -1.47 (112.93) | 10.40 (56.69) | -15.04 (161.72) | -59.66 (123.62)
  Cortisol: Change from week 0 to week 52 | 3.60 (50.63) | 7.54 (33.71) | -14.15 (43.84) | 21.67 (46.62) | -4.01 (47.82) | 12.59 (37.65)

89. Secondary Outcome: Change in Hormone Level: Dehydroepiandrosterone Sulfate (DHEAS) From Baseline at Week 16
Description: Change in DHEAS from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 11 | 13 | 5 | 31 | 16
umol/L | 0.16 (1.74) | 0.21 (0.95) | 0.25 (1.10) | 1.00 (1.42) | 0.20 (1.48) | 0.46 (1.13)

90. Secondary Outcome: Change in Hormone Level: Dehydroepiandrosterone Sulfate (DHEAS) From Baseline at Week 52
Description: Change in DHEAS from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 8 | 12 | 4 | 28 | 12
umol/L | 0.77 (1.18) | 0.76 (0.97) | 0.25 (0.66) | 0.74 (1.26) | 0.55 (1.01) | 0.76 (1.01)

91. Secondary Outcome: Change in Hormone Level: Luteinising Hormone (LH), Follicle Stimulating Hormone (FSH) From Baseline at Week 16
Description: Change in LH and FSH from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 12 | 13 | 7 | 30 | 19
IU/L
  LH: Change from week 0 to week 16 | -0.04 (1.28) | 0.06 (0.74) | -0.07 (0.25) | 0.22 (0.42) | -0.05 (0.97) | 0.12 (0.63)
  FSH: Change from week 0 to week 16: number analyzed (Participants) | 16 | 9 | 11 | 7 | 27 | 16
  FSH: Change from week 0 to week 16 | -0.2 (2.5) | 0.2 (1.0) | -0.1 (1.3) | 1.0 (1.1) | -0.2 (2.1) | 0.5 (1.1)

92. Secondary Outcome: Change in Hormone Level: Luteinising Hormone (LH), Follicle Stimulating Hormone (FSH) From Baseline at Week 52
Description: Change in LH and FSH from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 16 | 10 | 11 | 5 | 27 | 15
IU/L
  LH: Change from week 0 to week 52 | 0.16 (2.33) | 0.06 (0.79) | 0.37 (0.96) | 0.30 (0.51) | 0.24 (1.87) | 0.14 (0.70)
  FSH: Change from week 0 to week 52: number analyzed (Participants) | 12 | 7 | 11 | 5 | 23 | 12
  FSH: Change from week 0 to week 52 | 1.1 (3.9) | 0.4 (1.6) | 0.4 (1.8) | 0.7 (1.6) | 0.8 (3.1) | 0.6 (1.5)

93. Secondary Outcome: Change in Hormone Level: Estradiol (Females) From Baseline at Week 16
Description: Change in estradiol (only for females) from baseline to week 16 is presented.
Time Frame: Week 0, week 16
Population: SAS which included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = number of female participants who contributed to the analysis. Combined data of Part A and B for liraglutide and placebo was planned to be reported.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 9 | 4 | 6 | 2 | 15 | 6
picograms per milliliter (pg/mL) | 0.9 (15.8) | 9.2 (11.9) | 1.6 (3.8) | 0 (0) | 1.2 (12.2) | 6.1 (10.4)

94. Secondary Outcome: Change in Hormone Level: Estradiol (Females) From Baseline at Week 52
Description: Change in estradiol (only for females) from baseline to week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 93
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 7 | 4 | 8 | 1 | 15 | 5
pg/mL | 7.0 (32.6) | 13.7 (21.6) | 1.6 (4.5) | 0 (NA) — As there was only one participant evaluated for the Part B: Placebo arm; Mean and SD could not be calculated. | 4.1 (21.8) | 11.0 (19.7)

95. Secondary Outcome: Change in Hormone Level: Testosterone (Males) From Baseline at Week 16
Description: Change in testosterone (only for males) from baseline to week 16 is presented. The testosterone analysis for Part B could not be performed due to an unforeseen change in the assay used by the central laboratory to measure testosterone during the trial. This change in methodology prevented a direct comparison of values measured at different time points during the trial.
Time Frame: Week 0, week 16
Population: SAS which included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = number of male participants who contributed to the analysis.
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Part A: Liraglutide | Part A: Placebo
Number analyzed (Participants) | 8 | 7
nanomoles per liter (nmol/L) | 1.55 (2.01) | 0.61 (1.66)

96. Secondary Outcome: Change in Hormone Level: Testosterone (Males) From Baseline at Week 52
Description: Change in testosterone (only for males) from baseline to week 52 is presented. The testosterone analysis for Part B could not be performed due to an unforeseen change in the assay used by the central laboratory to measure testosterone during the trial. This change in methodology prevented a direct comparison of values measured at different time points during the trial.
Time Frame: Week 0, week 52
Population: as for outcome 95
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part A: Liraglutide | Part A: Placebo
Number analyzed (Participants) | 8 | 5
nmol/L | 0.62 (1.40) | -0.34 (1.51)

97. Secondary Outcome: Number of Participants With Change in Pubertal Status From Baseline at Week 16
Description: This outcome measure presents "pubertal status results" which is based on Tanner staging recorded at baseline (week 0), week 16. Tanner Stages is a scale that defines physical measurements of development based on external primary and secondary sex characteristics. It was used in this study to assess pubertal development with values ranging from Stage 1 (pre-pubertal characteristics) to Stage 5 (adult or mature characteristics). Results are presented for the following categories: 1) For female: breast development and pubic hair development, 2) For male: penis development and pubic hair development. Each category shows number of participants in stages 1 to 5, where stage 1 represents "early pubertal development" and stage 5 represents "pubertal development equivalent to that of an adult".
Time Frame: Week 0, week 16
Population: as for outcome 67
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 11 | 7 | 11 | 5 | 22 | 12
Participants
  Week 0: Breast development (for female): number analyzed (Participants) | 11 | 5 | 11 | 2 | 22 | 7
  Week 0: Breast development (for female): Stage 1 | 0 | 0 | 11 | 2 | 11 | 2
  Week 0: Breast development (for female): Stage 2 | 1 | 0 | 0 | 0 | 1 | 0
  Week 0: Breast development (for female): Stage 3 | 8 | 2 | 0 | 0 | 8 | 2
  Week 0: Breast development (for female): Stage 4 | 0 | 1 | 0 | 0 | 0 | 1
  Week 0: Breast development (for female): Stage 5 | 2 | 2 | 0 | 0 | 2 | 2
  Week 16: Breast development (for female): number analyzed (Participants) | 10 | 5 | 9 | 2 | 19 | 7
  Week 16: Breast development (for female): Stage 1 | 0 | 0 | 6 | 2 | 6 | 2
  Week 16: Breast development (for female): Stage 2 | 1 | 0 | 3 | 0 | 4 | 0
  Week 16: Breast development (for female): Stage 3 | 7 | 1 | 0 | 0 | 7 | 1
  Week 16: Breast development (for female): Stage 4 | 0 | 2 | 0 | 0 | 0 | 2
  Week 16: Breast development (for female): Stage 5 | 2 | 2 | 0 | 0 | 2 | 2
  Week 0: Pubic hair development (for female): number analyzed (Participants) | 11 | 5 | 11 | 2 | 22 | 7
  Week 0: Pubic hair development (for female): Stage 1 | 1 | 0 | 6 | 1 | 7 | 1
  Week 0: Pubic hair development (for female): Stage 2 | 2 | 0 | 3 | 0 | 5 | 0
  Week 0: Pubic hair development (for female): Stage 3 | 3 | 2 | 0 | 1 | 3 | 3
  Week 0: Pubic hair development (for female): Stage 4 | 3 | 1 | 2 | 0 | 5 | 1
  Week 0: Pubic hair development (for female): Stage 5 | 2 | 2 | 0 | 0 | 2 | 2
  Week 16: Pubic hair development (for female): number analyzed (Participants) | 10 | 5 | 9 | 2 | 19 | 7
  Week 16: Pubic hair development (for female): Stage 1 | 1 | 0 | 3 | 1 | 4 | 1
  Week 16: Pubic hair development (for female): Stage 2 | 1 | 0 | 5 | 0 | 6 | 0
  Week 16: Pubic hair development (for female): Stage 3 | 4 | 1 | 0 | 1 | 4 | 2
  Week 16: Pubic hair development (for female): Stage 4 | 2 | 2 | 1 | 0 | 3 | 2
  Week 16: Pubic hair development (for female): Stage 5 | 2 | 2 | 0 | 0 | 2 | 2
  Week 0: Pubic hair development (for male): number analyzed (Participants) | 9 | 7 | 6 | 5 | 15 | 12
  Week 0: Pubic hair development (for male): Stage 1 | 0 | 0 | 6 | 3 | 6 | 3
  Week 0: Pubic hair development (for male): Stage 2 | 3 | 0 | 0 | 1 | 3 | 1
  Week 0: Pubic hair development (for male): Stage 3 | 2 | 4 | 0 | 1 | 2 | 5
  Week 0: Pubic hair development (for male): Stage 4 | 2 | 2 | 0 | 0 | 2 | 2
  Week 0: Pubic hair development (for male): Stage 5 | 2 | 1 | 0 | 0 | 2 | 1
  Week 16: Pubic hair development (for male): number analyzed (Participants) | 9 | 7 | 6 | 5 | 15 | 12
  Week 16: Pubic hair development (for male): Stage 1 | 0 | 0 | 6 | 1 | 6 | 1
  Week 16: Pubic hair development (for male): Stage 2 | 2 | 0 | 0 | 3 | 2 | 3
  Week 16: Pubic hair development (for male): Stage 3 | 2 | 3 | 0 | 1 | 2 | 4
  Week 16: Pubic hair development (for male): Stage 4 | 2 | 2 | 0 | 0 | 2 | 2
  Week 16: Pubic hair development (for male): Stage 5 | 3 | 2 | 0 | 0 | 3 | 2
  Week 0: Penis development (for male): number analyzed (Participants) | 9 | 7 | 6 | 5 | 15 | 12
  Week 0: Penis development (for male): Stage 1 | 0 | 1 | 6 | 5 | 6 | 6
  Week 0: Penis development (for male): Stage 2 | 4 | 3 | 0 | 0 | 4 | 3
  Week 0: Penis development (for male): Stage 3 | 1 | 1 | 0 | 0 | 1 | 1
  Week 0: Penis development (for male): Stage 4 | 3 | 2 | 0 | 0 | 3 | 2
  Week 0: Penis development (for male): Stage 5 | 1 | 0 | 0 | 0 | 1 | 0
  Week 16: Penis development (for male): number analyzed (Participants) | 9 | 7 | 6 | 5 | 15 | 12
  Week 16: Penis development (for male): Stage 1 | 0 | 1 | 5 | 5 | 5 | 6
  Week 16: Penis development (for male): Stage 2 | 2 | 1 | 1 | 0 | 3 | 1
  Week 16: Penis development (for male): Stage 3 | 2 | 3 | 0 | 0 | 2 | 3
  Week 16: Penis development (for male): Stage 4 | 2 | 1 | 0 | 0 | 2 | 1
  Week 16: Penis development (for male): Stage 5 | 3 | 1 | 0 | 0 | 3 | 1

98. Secondary Outcome: Number of Participants With Change in Pubertal Status From Baseline at Week 52
Description: This outcome measure presents "pubertal status results" which is based on Tanner staging recorded at baseline (week 0) and week 52. Tanner Stages is a scale that defines physical measurements of development based on external primary and secondary sex characteristics. It was used in this study to assess pubertal development with values ranging from Stage 1 (pre-pubertal characteristics) to Stage 5 (adult or mature characteristics). Results are presented for the following categories: 1) For female: breast development and pubic hair development, 2) For male: penis development and pubic hair development. Each category shows number of participants in stages 1 to 5, where stage 1 represents "early pubertal development" and stage 5 represents "pubertal development equivalent to that of an adult".
Time Frame: Week 0, week 52
Population: as for outcome 67
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 11 | 7 | 11 | 5 | 22 | 12
Participants
  Week 0: Breast development (for female): number analyzed (Participants) | 11 | 5 | 11 | 2 | 22 | 7
  Week 0: Breast development (for female): Stage 1 | 0 | 0 | 11 | 2 | 11 | 2
  Week 0: Breast development (for female): Stage 2 | 1 | 0 | 0 | 0 | 1 | 0
  Week 0: Breast development (for female): Stage 3 | 8 | 2 | 0 | 0 | 8 | 2
  Week 0: Breast development (for female): Stage 4 | 0 | 1 | 0 | 0 | 0 | 1
  Week 0: Breast development (for female): Stage 5 | 2 | 2 | 0 | 0 | 2 | 2
  Week 52: Breast development (for female): number analyzed (Participants) | 9 | 5 | 8 | 1 | 17 | 6
  Week 52: Breast development (for female): Stage 1 | 0 | 0 | 2 | 1 | 2 | 1
  Week 52: Breast development (for female): Stage 2 | 0 | 0 | 4 | 0 | 4 | 0
  Week 52: Breast development (for female): Stage 3 | 5 | 1 | 2 | 0 | 7 | 1
  Week 52: Breast development (for female): Stage 4 | 1 | 2 | 0 | 0 | 1 | 2
  Week 52: Breast development (for female): Stage 5 | 3 | 2 | 0 | 0 | 3 | 2
  Week 0: Pubic hair development (for female): number analyzed (Participants) | 11 | 5 | 11 | 2 | 22 | 7
  Week 0: Pubic hair development (for female): Stage 1 | 1 | 0 | 6 | 1 | 7 | 1
  Week 0: Pubic hair development (for female): Stage 2 | 2 | 0 | 3 | 0 | 5 | 0
  Week 0: Pubic hair development (for female): Stage 3 | 3 | 2 | 0 | 1 | 3 | 3
  Week 0: Pubic hair development (for female): Stage 4 | 3 | 1 | 2 | 0 | 5 | 1
  Week 0: Pubic hair development (for female): Stage 5 | 2 | 2 | 0 | 0 | 2 | 2
  Week 52: Pubic hair development (for female): number analyzed (Participants) | 9 | 5 | 8 | 1 | 17 | 6
  Week 52: Pubic hair development (for female): Stage 1 | 1 | 0 | 1 | 0 | 2 | 0
  Week 52: Pubic hair development (for female): Stage 2 | 1 | 0 | 2 | 0 | 3 | 0
  Week 52: Pubic hair development (for female): Stage 3 | 2 | 1 | 4 | 1 | 6 | 2
  Week 52: Pubic hair development (for female): Stage 4 | 3 | 2 | 1 | 0 | 4 | 2
  Week 52: Pubic hair development (for female): Stage 5 | 2 | 2 | 0 | 0 | 2 | 2
  Week 0: Pubic hair development (for male): number analyzed (Participants) | 9 | 7 | 6 | 5 | 15 | 12
  Week 0: Pubic hair development (for male): Stage 1 | 0 | 0 | 6 | 3 | 6 | 3
  Week 0: Pubic hair development (for male): Stage 2 | 3 | 0 | 0 | 1 | 3 | 1
  Week 0: Pubic hair development (for male): Stage 3 | 2 | 4 | 0 | 1 | 2 | 5
  Week 0: Pubic hair development (for male): Stage 4 | 2 | 2 | 0 | 0 | 2 | 2
  Week 0: Pubic hair development (for male): Stage 5 | 2 | 1 | 0 | 0 | 2 | 1
  Week 52: Pubic hair development (for male): number analyzed (Participants) | 9 | 6 | 5 | 3 | 14 | 9
  Week 52: Pubic hair development (for male): Stage 1 | 0 | 0 | 4 | 0 | 4 | 0
  Week 52: Pubic hair development (for male): Stage 2 | 0 | 0 | 1 | 1 | 1 | 1
  Week 52: Pubic hair development (for male): Stage 3 | 3 | 2 | 0 | 1 | 3 | 3
  Week 52: Pubic hair development (for male): Stage 4 | 3 | 3 | 0 | 1 | 3 | 4
  Week 52: Pubic hair development (for male): Stage 5 | 3 | 1 | 0 | 0 | 3 | 1
  Week 0: Penis development (for male): number analyzed (Participants) | 9 | 7 | 6 | 5 | 15 | 12
  Week 0: Penis development (for male): Stage 1 | 0 | 1 | 6 | 5 | 6 | 6
  Week 0: Penis development (for male): Stage 2 | 4 | 3 | 0 | 0 | 4 | 3
  Week 0: Penis development (for male): Stage 3 | 1 | 1 | 0 | 0 | 1 | 1
  Week 0: Penis development (for male): Stage 4 | 3 | 2 | 0 | 0 | 3 | 2
  Week 0: Penis development (for male): Stage 5 | 1 | 0 | 0 | 0 | 1 | 0
  Week 52: Penis development (for male): number analyzed (Participants) | 9 | 6 | 5 | 3 | 14 | 9
  Week 52: Penis development (for male): Stage 1 | 0 | 1 | 3 | 2 | 3 | 3
  Week 52: Penis development (for male): Stage 2 | 1 | 1 | 2 | 1 | 3 | 2
  Week 52: Penis development (for male): Stage 3 | 2 | 1 | 0 | 0 | 2 | 1
  Week 52: Penis development (for male): Stage 4 | 3 | 2 | 0 | 0 | 3 | 2
  Week 52: Penis development (for male): Stage 5 | 3 | 1 | 0 | 0 | 3 | 1

99. Secondary Outcome: Number of Participants With Change in Physical Examination From Baseline at Week 16
Description: This outcome measure presents number of participants with physical examination findings, "normal; abnormal, not clinically significant (NCS) or abnormal, clinically significant (CS)" at baseline (week 0), week 16. These findings were categorised by the investigator. Results include examination of: general appearance; head, ears, eyes, nose, throat, neck; respiratory system; cardiovascular system (CVS); gastrointestinal (GI) system including mouth; musculoskeletal system; central nervous system (CNS) and peripheral nervous system (PNS); skin; thyroid gland and lymph node palpation.
Time Frame: Week 0, week 16
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 20 | 12 | 17 | 7 | 37 | 19
Participants
  General Appearance: Week 0: Normal | 14 | 10 | 12 | 5 | 26 | 15
  General Appearance: Week 0: Abnormal, NCS | 2 | 1 | 3 | 1 | 5 | 2
  General Appearance: Week 0: Abnormal, CS | 4 | 1 | 2 | 1 | 6 | 2
  General Appearance: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  General Appearance: Week 16: Normal | 14 | 11 | 11 | 5 | 25 | 16
  General Appearance: Week 16: Abnormal, NCS | 1 | 0 | 4 | 1 | 5 | 1
  General Appearance: Week 16: Abnormal, CS | 4 | 1 | 0 | 1 | 4 | 2
  Head, ears, eyes, nose, throat, neck: Week 0: Normal | 19 | 10 | 15 | 6 | 34 | 16
  Head, ears, eyes, nose, throat, neck: Week 0: Abnormal, NCS | 1 | 2 | 2 | 1 | 3 | 3
  Head, ears, eyes, nose, throat, neck: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Head, ears, eyes, nose, throat, neck: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  Head, ears, eyes, nose, throat, neck: Week 16: Normal | 18 | 12 | 15 | 7 | 33 | 19
  Head, ears, eyes, nose, throat, neck: Week 16: Abnormal, NCS | 1 | 0 | 0 | 0 | 1 | 0
  Head, ears, eyes, nose, throat, neck: Week 16: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory system: Week 0: Normal | 20 | 12 | 16 | 7 | 36 | 19
  Respiratory system: Week 0: Abnormal, NCS | 0 | 0 | 1 | 0 | 1 | 0
  Respiratory system: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory system: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  Respiratory system: Week 16: Normal | 19 | 12 | 15 | 7 | 34 | 19
  Respiratory system: Week 16: Abnormal, NCS | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory system: Week 16: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Cardiovascular system: Week 0: Normal | 19 | 12 | 17 | 7 | 36 | 19
  Cardiovascular system: Week 0: Abnormal, NCS | 1 | 0 | 0 | 0 | 1 | 0
  Cardiovascular system: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Cardiovascular system: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  Cardiovascular system: Week 16: Normal | 18 | 12 | 15 | 7 | 33 | 19
  Cardiovascular system: Week 16: Abnormal, NCS | 1 | 0 | 0 | 0 | 1 | 0
  Cardiovascular system: Week 16: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  GI system including mouth: Week 0: Normal | 19 | 12 | 17 | 7 | 36 | 19
  GI system including mouth: Week 0: Abnormal, NCS | 1 | 0 | 0 | 0 | 1 | 0
  GI system including mouth: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  GI system including mouth: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  GI system including mouth: Week 16: Normal | 17 | 12 | 15 | 7 | 32 | 19
  GI system including mouth: Week 16: Abnormal, NCS | 2 | 0 | 0 | 0 | 2 | 0
  GI system including mouth: Week 16: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal system: Week 0: Normal | 15 | 9 | 14 | 6 | 29 | 15
  Musculoskeletal system: Week 0: Abnormal, NCS | 3 | 2 | 3 | 1 | 6 | 3
  Musculoskeletal system: Week 0: Abnormal, CS | 2 | 1 | 0 | 0 | 2 | 1
  Musculoskeletal system: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  Musculoskeletal system: Week 16: Normal | 16 | 9 | 11 | 6 | 27 | 15
  Musculoskeletal system: Week 16: Abnormal, NCS | 2 | 1 | 4 | 1 | 6 | 2
  Musculoskeletal system: Week 16: Abnormal, CS | 1 | 2 | 0 | 0 | 1 | 2
  CNS and PNS: Week 0: Normal | 16 | 10 | 15 | 6 | 31 | 16
  CNS and PNS: Week 0: Abnormal, NCS | 2 | 0 | 1 | 1 | 3 | 1
  CNS and PNS: Week 0: Abnormal, CS | 2 | 2 | 1 | 0 | 3 | 2
  CNS and PNS: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  CNS and PNS: Week 16: Normal | 15 | 11 | 14 | 7 | 29 | 18
  CNS and PNS: Week 16: Abnormal, NCS | 2 | 0 | 1 | 0 | 3 | 0
  CNS and PNS: Week 16: Abnormal, CS | 2 | 1 | 0 | 0 | 2 | 1
  Skin: Week 0: Normal | 11 | 7 | 10 | 6 | 21 | 13
  Skin: Week 0: Abnormal, NCS | 6 | 4 | 6 | 1 | 12 | 5
  Skin: Week 0: Abnormal, CS | 3 | 1 | 1 | 0 | 4 | 1
  Skin: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  Skin: Week 16: Normal | 12 | 8 | 10 | 6 | 22 | 14
  Skin: Week 16: Abnormal, NCS | 5 | 3 | 5 | 0 | 10 | 3
  Skin: Week 16: Abnormal, CS | 2 | 1 | 0 | 1 | 2 | 2
  Thyroid gland: Week 0: Normal | 20 | 12 | 17 | 7 | 37 | 19
  Thyroid gland: Week 0: Abnormal, NCS | 0 | 0 | 0 | 0 | 0 | 0
  Thyroid gland: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Thyroid gland: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  Thyroid gland: Week 16: Normal | 19 | 12 | 15 | 7 | 34 | 19
  Thyroid gland: Week 16: Abnormal, NCS | 0 | 0 | 0 | 0 | 0 | 0
  Thyroid gland: Week 16: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Lymph node palpation: Week 0: Normal | 19 | 12 | 17 | 7 | 36 | 19
  Lymph node palpation: Week 0: Abnormal, NCS | 1 | 0 | 0 | 0 | 1 | 0
  Lymph node palpation: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Lymph node palpation: Week 16: number analyzed (Participants) | 19 | 12 | 15 | 7 | 34 | 19
  Lymph node palpation: Week 16: Normal | 19 | 12 | 15 | 7 | 34 | 19
  Lymph node palpation: Week 16: Abnormal, NCS | 0 | 0 | 0 | 0 | 0 | 0
  Lymph node palpation: Week 16: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0

100. Secondary Outcome: Number of Participants With Change in Physical Examination From Baseline at Week 52
Description: This outcome measure presents number of participants with physical examination findings, "normal; abnormal, not clinically significant (NCS) or abnormal, clinically significant (CS)" at baseline (week 0) and week 52. These findings were categorised by the investigator. Results include examination of: general appearance; head, ears, eyes, nose, throat, neck; respiratory system; cardiovascular system (CVS); gastrointestinal (GI) system including mouth; musculoskeletal system; central nervous system (CNS) and peripheral nervous system (PNS); skin; thyroid gland and lymph node palpation.
Time Frame: Week 0, week 52
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 20 | 12 | 17 | 7 | 37 | 19
Participants
  General Appearance: Week 0: Normal | 14 | 10 | 12 | 5 | 26 | 15
  General Appearance: Week 0: Abnormal, NCS | 2 | 1 | 3 | 1 | 5 | 2
  General Appearance: Week 0: Abnormal, CS | 4 | 1 | 2 | 1 | 6 | 2
  General Appearance: Week 52: number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
  General Appearance: Week 52: Normal | 13 | 10 | 9 | 5 | 22 | 15
  General Appearance: Week 52: Abnormal, NCS | 1 | 0 | 2 | 0 | 3 | 0
  General Appearance: Week 52: Abnormal, CS | 3 | 1 | 1 | 0 | 4 | 1
  Head, ears, eyes, nose, throat, neck: Week 0: Normal | 19 | 10 | 15 | 6 | 34 | 16
  Head, ears, eyes, nose, throat, neck: Week 0: Abnormal, NCS | 1 | 2 | 2 | 1 | 3 | 3
  Head, ears, eyes, nose, throat, neck: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Head, ears, eyes, nose, throat, neck: Week 52: number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
  Head, ears, eyes, nose, throat, neck: Week 52: Normal | 15 | 11 | 12 | 4 | 27 | 15
  Head, ears, eyes, nose, throat, neck: Week 52: Abnormal, NCS | 2 | 0 | 0 | 1 | 2 | 1
  Head, ears, eyes, nose, throat, neck: Week 52: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory system: Week 0: Normal | 20 | 12 | 16 | 7 | 36 | 19
  Respiratory system: Week 0: Abnormal, NCS | 0 | 0 | 1 | 0 | 1 | 0
  Respiratory system: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Cardiovascular system: Week 0: Normal | 19 | 12 | 17 | 7 | 36 | 19
  Cardiovascular system: Week 0: Abnormal, NCS | 1 | 0 | 0 | 0 | 1 | 0
  Cardiovascular system: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Cardiovascular system: Week 52: number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
  Cardiovascular system: Week 52: Normal | 17 | 10 | 12 | 5 | 29 | 15
  Cardiovascular system: Week 52: Abnormal, NCS | 0 | 0 | 0 | 0 | 0 | 0
  Cardiovascular system: Week 52: Abnormal, CS | 0 | 1 | 0 | 0 | 0 | 1
  GI system including mouth: Week 0: Normal | 19 | 12 | 17 | 7 | 36 | 19
  GI system including mouth: Week 0: Abnormal, NCS | 1 | 0 | 0 | 0 | 1 | 0
  GI system including mouth: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  GI system including mouth: Week 52: number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
  GI system including mouth: Week 52: Normal | 16 | 11 | 12 | 5 | 28 | 16
  GI system including mouth: Week 52: Abnormal, NCS | 1 | 0 | 0 | 0 | 1 | 0
  GI system including mouth: Week 52: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal system: Week 0: Normal | 15 | 9 | 14 | 6 | 29 | 15
  Musculoskeletal system: Week 0: Abnormal, NCS | 3 | 2 | 3 | 1 | 6 | 3
  Musculoskeletal system: Week 0: Abnormal, CS | 2 | 1 | 0 | 0 | 2 | 1
  Musculoskeletal system: Week 52: number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
  Musculoskeletal system: Week 52: Normal | 15 | 10 | 10 | 5 | 25 | 15
  Musculoskeletal system: Week 52: Abnormal, NCS | 1 | 1 | 2 | 0 | 3 | 1
  Musculoskeletal system: Week 52: Abnormal, CS | 1 | 0 | 0 | 0 | 1 | 0
  CNS and PNS: Week 0: Normal | 16 | 10 | 15 | 6 | 31 | 16
  CNS and PNS: Week 0: Abnormal, NCS | 2 | 0 | 1 | 1 | 3 | 1
  CNS and PNS: Week 0: Abnormal, CS | 2 | 2 | 1 | 0 | 3 | 2
  CNS and PNS: Week 52: number analyzed (Participants) | 16 | 11 | 12 | 5 | 28 | 16
  CNS and PNS: Week 52: Normal | 13 | 10 | 11 | 4 | 24 | 14
  CNS and PNS: Week 52: Abnormal, NCS | 1 | 0 | 0 | 1 | 1 | 1
  CNS and PNS: Week 52: Abnormal, CS | 2 | 1 | 1 | 0 | 3 | 1
  Skin: Week 0: Normal | 11 | 7 | 10 | 6 | 21 | 13
  Skin: Week 0: Abnormal, NCS | 6 | 4 | 6 | 1 | 12 | 5
  Skin: Week 0: Abnormal, CS | 3 | 1 | 1 | 0 | 4 | 1
  Skin: Week 52: number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
  Skin: Week 52: Normal | 13 | 8 | 9 | 4 | 22 | 12
  Skin: Week 52: Abnormal, NCS | 3 | 2 | 3 | 0 | 6 | 2
  Skin: Week 52: Abnormal, CS | 1 | 1 | 0 | 1 | 1 | 2
  Thyroid gland: Week 0: Normal | 20 | 12 | 17 | 7 | 37 | 19
  Thyroid gland: Week 0: Abnormal, NCS | 0 | 0 | 0 | 0 | 0 | 0
  Thyroid gland: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Thyroid gland: Week 52: number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
  Thyroid gland: Week 52: Normal | 17 | 11 | 12 | 5 | 29 | 16
  Thyroid gland: Week 52: Abnormal, NCS | 0 | 0 | 0 | 0 | 0 | 0
  Thyroid gland: Week 52: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Lymph node palpation: Week 0: Normal | 19 | 12 | 17 | 7 | 36 | 19
  Lymph node palpation: Week 0: Abnormal, NCS | 1 | 0 | 0 | 0 | 1 | 0
  Lymph node palpation: Week 0: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0
  Lymph node palpation: Week 52: number analyzed (Participants) | 17 | 11 | 12 | 5 | 29 | 16
  Lymph node palpation: Week 52: Normal | 17 | 11 | 12 | 5 | 29 | 16
  Lymph node palpation: Week 52: Abnormal, NCS | 0 | 0 | 0 | 0 | 0 | 0
  Lymph node palpation: Week 52: Abnormal, CS | 0 | 0 | 0 | 0 | 0 | 0

101. Secondary Outcome: Height Velocity at Week 16
Description: Height velocity was the change in height per year. The height velocity was calculated as the difference between current height and baseline divided by by time duration in days between those measurement time points and multiplied by 365 days. Height velocity calculated at Weeks 16 is presented.
Time Frame: Week 16
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: Centimeters/year (cm/yr)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 18 | 12 | 16 | 7 | 34 | 19
Centimeters/year (cm/yr) | 2.113 (3.084) | 2.718 (4.281) | 4.190 (2.604) | 6.898 (2.886) | 3.090 (3.014) | 4.258 (4.274)

102. Secondary Outcome: Height Velocity at Week 52
Description: Height velocity was the change in height per year. The height velocity was calculated as the difference between current height and baseline divided by by time duration in days between those measurement time points and multiplied by 365 days. Height velocity calculated at Week 52 are presented.
Time Frame: week 52
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: Centimeters/year (cm/yr)
Arm/Group | Part A: Liraglutide | Part A: Placebo | Part B: Liraglutide | Part B: Placebo | Part A+B: Liraglutide | Part A+B: Placebo
Number analyzed (Participants) | 17 | 11 | 14 | 6 | 31 | 17
Centimeters/year (cm/yr) | 1.564 (1.285) | 1.839 (1.658) | 4.752 (2.250) | 5.620 (1.690) | 3.004 (2.383) | 3.173 (2.466)

103. Secondary Outcome: Part A: Number of Participants With Change in Columbia Suicidality Severity Rating Scale (C-SSRS) at Week 16
Description: C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess suicidality, suicidal behaviour, suicidal ideation. Suicidality: emergence of any suicidal ideation or suicidal behaviour. Suicidal behaviour: when response is "yes" for any of the questions- actual attempt to suicide, engaged in non-suicidal self-injurious behaviour, interrupted attempt, aborted attempt, preparatory acts. Suicidal ideation: when response is "yes" for any of the questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide. This outcome measure presents number of participants with "suicidal ideation or suicidal behaviour on C-SSRS" assessed at baseline (week 0), week 16. The questionnaire was not used in Part B due to the young age of the participants in Part B.
Time Frame: Week 0, week 16
Population: SAS which included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = number of participants who contributed to the analysis. Number Analyzed = number of participants with available data. This outcome measure was planned to be analyzed for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo
Number analyzed (Participants) | 20 | 12
Participants
  Week 0: Suicidal ideation | 1 | 3
  Week 0: Suicidal behaviour | 0 | 0
  Week 16: Suicidal ideation: number analyzed (Participants) | 19 | 12
  Week 16: Suicidal ideation | 1 | 1
  Week 16: Suicidal behaviour: number analyzed (Participants) | 18 | 12
  Week 16: Suicidal behaviour | 0 | 0

104. Secondary Outcome: Part A: Number of Participants With Change in Columbia Suicidality Severity Rating Scale (C-SSRS) at Week 52
Description: C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess suicidality, suicidal behaviour, suicidal ideation. Suicidality: emergence of any suicidal ideation or suicidal behaviour. Suicidal behaviour: when response is "yes" for any of the questions- actual attempt to suicide, engaged in non-suicidal self-injurious behaviour, interrupted attempt, aborted attempt, preparatory acts. Suicidal ideation: when response is "yes" for any of the questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide. This outcome measure presents number of participants with "suicidal ideation or suicidal behaviour on C-SSRS" assessed at baseline (week 0), week 52. The questionnaire was not used in Part B due to the young age of the participants in Part B.
Time Frame: Week 0, week 52
Population: as for outcome 103
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Liraglutide | Part A: Placebo
Number analyzed (Participants) | 20 | 12
Participants
  Week 0: Suicidal ideation | 1 | 3
  Week 0: Suicidal behaviour | 0 | 0
  Week 52: Suicidal ideation: number analyzed (Participants) | 18 | 11
  Week 52: Suicidal ideation | 1 | 0
  Week 52: Suicidal behaviour: number analyzed (Participants) | 18 | 11
  Week 52: Suicidal behaviour | 0 | 0

105. Secondary Outcome: Part A: Change in Patient Reported Health Questionnaire-9 (PHQ-9) From Baseline at Week 16
Description: Change in Patient Health Questionnaire 9 (PHQ-9) was evaluated from baseline (week 0) to weeks 16. The PHQ-9 questionnaire is a 9-item depression module included in the patient health questionnaire, a self-administered diagnostic tool used for assessment of mental disorders. The PHQ-9 total score ranges from 0-27; total scores of 1-4 represent no depression, total scores of 5-9 represent mild depression, total scores of 10-14 represent moderate depression, total scores of 15-19 represent moderately severe depression and total scores of 20-27 represent severe depression. The questionnaire was not used in Part B due to the young age of the participants in Part B.
Time Frame: Week 0, week 16
Population: SAS which included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed = number of participants who contributed to the analysis. This outcome measure was planned to be analyzed for Part A only.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part A: Liraglutide | Part A: Placebo
Number analyzed (Participants) | 19 | 12
Score on a scale | -2 (4) | 1 (5)

106. Secondary Outcome: Part A: Change in Patient Reported Health Questionnaire-9 (PHQ-9) From Baseline at Week 52
Description: Change in Patient Health Questionnaire 9 (PHQ-9) was evaluated from baseline (week 0) to weeks 52. The PHQ-9 questionnaire is a 9-item depression module included in the patient health questionnaire, a self-administered diagnostic tool used for assessment of mental disorders. The PHQ-9 total score ranges from 0-27; total scores of 1-4 represent no depression, total scores of 5-9 represent mild depression, total scores of 10-14 represent moderate depression, total scores of 15-19 represent moderately severe depression and total scores of 20-27 represent severe depression. The questionnaire was not used in Part B due to the young age of the participants in Part B.
Time Frame: Week 0, week 52
Population: as for outcome 105
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part A: Liraglutide | Part A: Placebo
Number analyzed (Participants) | 18 | 11
Score on a scale | -2 (3) | 0 (3)

ADVERSE EVENTS:
Time Frame: From week 0 to week 54 Results are based on SAS which included all participants exposed to at least one dose of trial product. All AEs reported here are TEAEs. TEAE is as an event that had onset date during on-treatment period.
Description: On-treatment period: included AEs with onset date on or after first day of trial product administration; any of following dates, whichever came first: a) 14 days after last day on trial product, or b) Follow-up visit (week54) for participants with trial product discontinuation or c) Last study visit (participants withdrawn without follow-up visit (week 54)).
Arm/Group | Part A: Liraglutide | Part B: Liraglutide | Part A: Placebo | Part B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17 | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/20 | 2/17 | 0/12 | 1/7
Other Adverse Events (participants affected / at risk) | 16/20 | 17/17 | 10/12 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Liraglutide (N=20) | Part B: Liraglutide (N=17) | Part A: Placebo (N=12) | Part B: Placebo (N=7)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Liraglutide (N=20) | Part B: Liraglutide (N=17) | Part A: Placebo (N=12) | Part B: Placebo (N=7)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (8) | 3 (12) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (7) | 0 (0) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcitonin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood insulin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (30) | 7 (62) | 2 (4) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection viral (Infections and infestations) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear tube insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (4) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (8) | 2 (3) | 3 (6) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (4) | 2 (2) | 1 (2) | 2 (3)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insulin resistance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insulin-like growth factor decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (5) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overflow diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain prophylaxis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Precocious puberty (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroxine free decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 3 (4) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT02527200/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT02527200/SAP_001.pdf